CLINICAL TRIAL: NCT03905395
Title: Meditation and Mindfulness for Recurrent Pregnancy Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henriette Svarre Nielsen, MD, DMSc (Other)
Responsible Party: Sponsor-Investigator, Henriette Svarre Nielsen, MD, DMSc, Henriette Svarre Nielsen, MD, DMSc, Consultant, Head of Recurrent Pregnancy Loss Unit, Associate Professor, Rigshospitalet, Denmark, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-18038456
Record Dates: First submitted 2019-04-02; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Recurrent Pregnancy Loss
Keywords: Meditation; mindfulness; pregnancy loss; stress
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: A randomized trial where women in an experimental arm will receive 3 times a three hour work shop with introduction to meditation and mindfulness during a 7 week period. Women in the other arm will have no intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation and mindfulness intervention (Active Comparator): Women in the intervention arm will 3 times receive a three hours work shop with introduction to meditation and mindfulness over a 7 week period from a certified meditation instructor. Questionnaires before and after the intervention.
  Interventions: Behavioral: Meditation and mindfulness
- Control group (No Intervention): Women in the no intervention arm will receive no introduction to meditation and mindfulness - only questionnaires at the same time as the intervention group receives questionnaires.

INTERVENTIONS:
Behavioral: Meditation and mindfulness — Women in the intervention arm will 3 times receive a three hours work shop with introduction to meditation and mindfulness over a 7 week period from a certified meditation instructor. Questionnaires before and after the intervention.
  Arms: Meditation and mindfulness intervention

SUMMARY:
In the Danish Recurrent Pregnancy Loss Unit in Rigshospitalet in Copenhagen recurrent pregnancy loss (RPL) is defined as three og more consecutive pregnancy losses in accordance with current European guidelines.

RPL affects approximately 3% of couples trying to achieve parenthood. Most cases of RPL are unexplained and have no effective treatment to improve the chance of a live birth.

42% of the women referred to RPL Unit in Rigshospitalet has a high stress level where as it's 22% in the background population trying to achieve parenthood. It's also known that 8,8 % of RPL patients have a depression at referral where as it's 2,2 % in the background population trying to achieve parenthood.

The study is a RCT including 62 patients - 31 in each arm. One arm will be taught in meditation and mindfulness three courses over a 7 week period. This group will also do meditation every day for 7 weeks. The other arm will have no intervention.

This study will investigate if a 7 weeks course in meditation and mindfulness is a useful tool to reduce stress and the psychological consequences for women and their partner treated in RPL Unit in Rigshospitalet, Copenhagen. Furthermore this study will investigate if there's a marital benefit such as reinforcement in their relationsship from practicing meditation and mindfulness.

There is no previous study that has investigated meditation and mindfulness for RPL.

This study has the potential to establish mental health support as a supplement to the medical and clinical treatment for RPL patients.

DETAILED DESCRIPTION:
The loss of a desired pregnancy is a significant negative life event associated with grief comparable to the grief after a peri- or neonatal death. Recurrent pregnancy loss (RPL) defined as 3 or more pregnancy losses affects approximately 3% of couples trying to have children. Most cases of RPL are unexplained and have no effective treatment to improve the chance of a live birth.

42% of the women referred to RPL Unit in Rigshospitalet has a high stress level where as it's 22% in the background population trying to achieve parenthood. It's also known that 8,8% of RPL patients have a depression at referral where as it's 2,2 % in the background population trying to achieve parenthood.

This study will investigate if a 7 weeks course in meditation and mindfulness is a useful tool to reduce stress and the psychological consequences for women and their partner treated in RPL Unit in Rigshospitalet, Copenhagen.

Furthermore this study will investigate if there's a marital benefit from practicing meditation and mindfulness. The investigators will use four different scales to measure the participants stress, depression, marital benefit and fertility stress. Also the investigators will measure the participants before and after the intervention and 12 months after.

All participants will have to complete:

1. Major Depression Index, a validated self-rating depression scale, which is used both clinically and in epidemiological studie. The 6-point Likert scale ranges from 0 (no depression) to 50 (extreme depression).
2. Perceived Stress Scale, which is a validated 10-item-self-reporting scale for stress symptoms. The 5 point Likert scale ranges from 0 (no stress) to 40 (extreme stress).
3. The COMPI Fertility Problem Stress Scale, a validated scale measuring the impact of RPL on the woman and her interpersonal relationships.
4. The COMPI Marital Benefit Scale measuring if RPL has reinforced the couples mariage/relationship.

The investigators assume that meditation and mindfulness can improve the quality of life for the RPL patients and their coping strategies. It's the investigators purpose to contribute with new knowledge in this area for current and future patients.

The RPL Unit in Rigshospitalet doesn't have any psychological support apart from ordinary attention from the nurses. This study has the potential to establish mental health support as a supplement to the medical and clinical treatment for RPL patients, which is in high demand.

ELIGIBILITY:
Inclusion Criteria:

* Women with RPL
* Speaking, reading and understanding Danish
* Have given a written consent
* Have a male partner
* Have a stress score > 16 points on Perceived Stress Scale

Exclusion Criteria:

* If the patient is pregnant on inclusion day
* If the patient already is practing meditation and mindfulness
* If the patient has a depression
* If the patient develops a depression after inclusion in either arm

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Based on biological sex
Enrollment: 64 (Estimated)
Dates: Start 2019-02-02 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | 7 weeks
  Change from baseline to 7 weeks after date of first course day measured by Perceived Stress Scale. PSS is a validated 10-item-self-reporting scale for stress symptoms. The 5 point Likert scale ranges from 0 (no stress) to 40 (extreme stress). The higher score the more stress.
Perceived Stress Scale (PSS) | 12 months
  Change from baseline to 12 months after date of first course day measured by the Perceived Stress Scale. PSS is a validated 10-item-self-reporting scale for stress symptoms. The 5 point Likert scale ranges from 0 (no stress) to 40 (extreme stress). The higher score the more stress.

SECONDARY OUTCOMES:
COMPI Fertility Problem Stress Scale | 7 weeks
  Change from baseline to 7 weeks after date of first course day using the COMPI Fertility Problem Stress Scale.
  The COMPI Fertility Problem Stress Scale is a validated scale measuring the impact of RPL on the woman and her interpersonal relationships. Two questions asking if the experience of RPL has been stressful for the woman with five answering options. Followed by seven sub questions asking how big a load RPL has been for the patients interpersonal life with four answering options. The lower the score the higher stress.
Marital Benefit Scale | 7 weeks
  Change in marital benefit from baseline to 7 weeks after date of first course day using the COMPI Marital Benefit Scale.
  The COMPI Marital Benefit Scale has two questions asking what the RPL have mattered for their relationship/mariage:
  Five options to answer: totally disagree, partly disagree, neither agree or disagree, partly agree, totally agree. Answering "Totally agree" on both questions is defined as a high marital benefit.
COMPI Fertility Problem Stress Scale | 12 months
  Change in fertility problem stress from baseline to 12 months after date of first course day using the COMPI Fertility Problem Stress Scale.
  The COMPI Fertility Problem Stress Scale is a validated scale measuring the impact of RPL on the woman and her interpersonal relationships. Two questions used to assess how big a impact RPL has for the patient with five answering options. Followed by seven sub questions asking how big a load RPL has been for the patients interpersonal life with four answering options. The lower the score the higher stress.
Marital Benefit | 12 months
  Change in marital benefit from baseline to 12 months after date of first course day using the COMPI Marital Benefit Scale.
  The COMPI Marital Benefit Scale has two questions asking what the RPL have mattered for their relationship/mariage:
  Five options to answer: totally disagree, partly disagree, neither agree or disagree, partly agree, totally agree. Answering "Totally agree" on both questions is defined as a high marital benefit.
Major Depression Index (MDI) | 12 months
  Change in depression score from baseline to 12 months after date of first course day. Major Depression Index is a validated self-rating depression scale, which is used both clinically and in epidemiological studie. The 6-point Likert scale ranges from 0 (no depression) to 50 (extreme depression).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Kirchheiner Jensen, Nurse, Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Østerbro, Denmark

IPD SHARING:
Plan to Share IPD: No